CLINICAL TRIAL: NCT05605496
Title: A Multicenter, Open-label, Proof of Concept Phase II Aiming to Assess the Clinical and Biological Activity of Anti-netrin-1 (NP137) as Add on Therapy in Patients With Advanced/Metastatic Solid Tumors Treated by Standard Immunotherapies
Brief Title: NP137 Clinical and Biological Activities Assessment in Patients With Advanced/Metastatic Solid Tumors Treated by Standard Anti PD-1/PD-L1 Immunotherapies
Acronym: IMMUNONET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: NETRIS Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET21-296; EU number (Other: 2022-500634-28-00)
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors; Metastatic Solid Tumors
Keywords: Solid Tumors; NP137; anti-PD1/PDL1; Stable disease; Primary refractory; Secondary Refractory; Netrin-1; monoclonal antibody
MeSH Terms: interventions — netrin-1 inhibitor NP137

STUDY DESIGN:
Intervention Model Description: The 3 cohorts of patients will be conducted and analyzed independently. The sample size calculation will use an adaptive Simon 2-stage design based on the strategy developed by Lin and Shih (Biometrics 2004). This method allows checking the result at the first stage, adjusting the power and success rate if necessary, and adapting the decision rule accordingly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stable Disease (Experimental): Patients with a radiological documentation of SD according to RECIST V1.1 criteria following at least 12 weeks under standard PD-1/PD-L1 therapy. The initial evidence of SD is to be confirmed by a second assessment, no less than 4 weeks from the date of the first documented SD. Note : This treatment arm closed on 27/09/2024 due to non-feasibility.
  Interventions: Drug: NP137; Drug: anti-PD-1/PD-L1
- Primary refractory (Experimental): Patients with documented radiological PD or short-term SD (< 6months) according to RECIST V1.1 but with clinical benefit under PD-1/PD-L1 standard therapy.
  Interventions: Drug: NP137; Drug: anti-PD-1/PD-L1
- Secondary refractory (Experimental): Patients with documented radiological PD following an initial Objective Response or long-term SD (i.e. ≥6 months) according to RECIST V1.1, with clinical benefit under standard PD-1/PD-L1.
  Interventions: Drug: NP137; Drug: anti-PD-1/PD-L1

INTERVENTIONS:
Drug: NP137 — IV infusion, 14mg/kg, Q3W
Drug: anti-PD-1/PD-L1 — IV infusion, Q3W or Q6W anti-PD1/PDL1 are standard treatments and are prepared and administred as per respective SmPC and institutional practice.

SUMMARY:
This study is a multicenter, open-label, proof-of-concept study aiming to assess the clinical and biological impact of NP137 when added to standard PD-1/PD-L1 blockade therapy in 3 independent cohorts of advanced or metastatic solid tumors with various sensitivity to anti-PD-1/PD-L1:

* Cohort 1 [Stable Disease]: Patients with a radiological documentation of SD according to RECIST V1.1 criteria following at least 12 weeks under standard anti PD-1/PD-L1 therapy. Note: This treatment arm closed on 27/09/2024 due to non-feasibility.
* Cohort 2 [primary refractory]: Patients with documented radiological PD or short-term SD (< 6months) according to RECIST V1.1 but with clinical benefit under PD-1/PD-L1 standard therapy.
* Cohort 3 [secondary refractory]: Patients with documented radiological PD following an initial Objective Response or long-term SD (i.e. ≥6 months) according to RECIST V1.1, with clinical benefit under standard PD-1/PD-L1.

DETAILED DESCRIPTION:
To be eligible to cohort 1 [stable disease], the initial evidence of SD is to be confirmed by a second assessment, no less than 4 weeks from the date of the first documented SD. To be eligible to cohorts 2 and 3 [primary and secondary refractory patients], patients must meet all the following criteria:

* Evidence of clinical benefit according to investigator assessment. The assessment of clinical benefit should be balanced by clinical judgment as to whether the patient is clinically deteriorating and unlikely to receive any benefit from continued anti-PD-1/PD-L1 treatment.
* Absence of symptoms and signs (including laboratory values, such as new or worsening hypercalcemia) indicating unequivocal progression of disease,
* Absence of decline in ECOG PS that can be attributed to disease progression,
* Absence of tumor progression at critical anatomical sites (e.g., leptomeningeal disease) that cannot be managed by protocol-allowed medical interventions.
* No ongoing clinically significant AE related to anti-PD-1/PD-L1.

During this study:

* All patients will receive NP137 (14 mg/kg, IV, Q3W) as add-on treatment to their standard anti-PD1 or anti-PDL1 treatment administered.
* To facilitate the study treatments administration and to not over burden patients, the study drug NP137 which is administered every 3 weeks (Q3W) will be associated to standard PD-1/PD-L1 therapies for which dosing are administered every 3 weeks or every 6 weeks (Q3W or Q6W). A treatment delay of up to 3 days is allowed before the start of a new cycle.

ELIGIBILITY:
Inclusion Criteria:

I1. Male or female patients aged ≥ 18 years at time of inform consent signature.

I2. Patient with histologically confirmed locally advanced / metastatic solid tumors of any histological types

I3. Patients treated with standard anti-PD-1/PD-L1 (e.g. pembrolizumab, atezolizumab, or any other ICI to be approved and reimbursed in France during the course of this trial, with a Q3W or Q6W schedule, either as monotherapy or in combination with chemotherapies according to their approved label). A positive list of eligible solid tumour types together with the associated anti-PD-1/PD-L1 standard therapy approved for each indication is provided in appendix 7. For any pathology not listed in this appendix but for which an anti-PD-1/PD-L1 has newly obtained a MA and is now reiumbursed in France, please refer to the section 0 of this protocol) and meet the following criteria :

* I3a. Cohort 1: Patient with RECIST 1.1.-defined SD under at least 12 weeks anti-PD-1/PD-L1. The initial evidence of SD is to be confirmed by a second assessment, no less than 4 weeks from the date of the first documented SD. Stable disease must be the best response observed since initiation of anti-PD-1/PD-L1 standard therapy or induction phase.
* I3b. Cohort 2: Patient with RECIST 1.1-defined PD under anti-PD-1/PD-L1 or short-term SD i.e. < 6 months as best response under anti-PD-1/PD-L1.
* I3c. Cohort 3: Patients with RECIST 1.1-defined PD under anti-PD1/PD-L1 after initial objective response (CR or PR) or long-term benefit i.e. SD lasting at least 6 months as per RECIST V1.1

Note 1 : For patients treated with an anti-PD-1/ PD-L1 previously combined to another anti-cancer agents of any type (including but not limited to chemotherapy/ other immunotherapy/ biological -or targeted agents) theseagents must be stopped 2 weeks or 5* t ½ whichever is shorter before C1D1 while anti-PD1 or anti PDL1 is continued according to Market Authorisation.

Note 2: Patients may have received a line of chemotherapy or any other standard anti-cancer agent after PD under anti-PD-1/PD-L1 but recurrence/progression under aPD-1/aPD-L1 y must have been documented ≤ 12 months before inclusion. Intercurrent chemotherapy or other standard agents must be stopped 2 weeks or 5* t ½ whichever is shorter before C1D1. Those patients will be then recruited in one of the refractory cohorts and could re-start an anti-PD1/PD-PL1 immediately in combination with NP137 at inclusion.

I4. Refractory cohorts: To be eligible in these cohorts, patients must meet all the following criteria:

* Evidence of clinical benefit according to investigator assessment. The assessment of clinical benefit should be balanced by clinical judgment as to whether the patient is clinically deteriorating and unlikely to receive any benefit from continued ICI treatment.
* Absence of symptoms and signs (including laboratory values, such as new or worsening hypercalcemia) indicating unequivocal progression of disease,
* Absence of decline in ECOG PS that can be attributed to disease progression,
* Absence of tumor progression at critical anatomical sites (e.g., leptomeningeal disease) that cannot be managed by protocol-allowed medical interventions.
* No ongoing clinically significant AE related to ICI.

I5. Patient with of at least one lesion measurable and evaluable as per RECIST V1.1 according to central imaging review before C1D1. Tumour lesions located in a previously irradiated area, or in an area subjected to other locoregional therapy, cannot be considered as measurable/evlaluable unless there has been a documentation of progression in the lesion.

I6. Availability of a representative archival tumor sample in formalin-fixed paraffin embedded (FFPE) block (primary tumor or metastasis) or newly obtained core or excisional biopsy of a tumor lesion together with an associated pathology report.

I7. Presence of at least one tumor lesion with a diameter ≥10 mm (≥20mm in case of a single biospsiable and RECIST 1.1 target lesion) visible by medical imaging and accessible to repeatable percutaneous sampling that permits core needle biopsy without unacceptable risk of a significant procedural complications, and suitable for retrieval of 4 cores using a 16-gauge diameter needle or larger.

Note: lesions to be biopsied should not be selected as RECIST target lesions unless there are no other lesions suitable for biopsy. If a RECIST target lesion is used for biopsy, the lesion must be ≥ 2 cm in longest diameter. Bone lesions are not adequate lesions for biopsies. Osteolytic lesions with soft tissue involvement cannot be biopsied.

I8. Life expectancy ≥ 3 months. I9. Eastern Cooperative Oncology Group performance status 0 or 1

I10. Demonstrate adequate cardiovascular function:

* QTcF < 470ms
* Resting BP systolic < 160mmHg and diastolic < 100mmHg
* LVEF > 50% as determined by transthoracic echocardiogram.

I11. Demonstrate adequate organ function as defined in table below, all screening laboratory tests should be performed within 7 days prior C1D1:

- Hematological : Absolute neutrophil count (ANC) ≥ 1.5 G/L (1500/µL)

Platelets ≥ 100 G/L (100000/µL) (transfusion within 21 days before C1D1 is allowed).

Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L-1 Packed red blood cell(pRBC) transfusion is allowed within past 2 weeks. Patient can be on stable dose of erythropoietin (≥3 months)

- Renal : Serum creatinine OR Creatinine clearance according to CKD-EPI (Appendix 3) ≤ 1.5 X upper limit of normal (ULN) OR ≥ 30 mL/min/1.73m2 for patient with creatinine levels > 1.5 ULN

- Hepatic : Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN

AST and ALT ≤ 2.5 X ULN (up to 5 ULN in case of liver metastases)

- Coagulation : International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN Note: This is applicable only for patients not receiving an anticoagulant treatment: patients receiving therapeutic anticoagulation must be on stable dose.

I12. Women of child-bearing potential must have a negative urine pregnancy test at screening (within 72 hours prior C1D1) and must agree to use 2 effective forms of contraception from the time of the treatment period and of the negative pregnancy test up 6 months after the end of their treatment. Effective forms of contraception are listing in Appendix 4.

I13. Fertile males must use a highly effective contraception during dosing period and through 3 months after final dose of study treatments.

I14. Patient should be able and willing to comply with study visits and procedures as per protocol.

I15. Patient should understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures performed.

I16. Patients must be covered by a medical insurance.

Exclusion Criteria:

E1. Patients eligible to curative treatment E2. For refractory cohorts: patients eligible to standard treatment with documented proof of activity in the tumor type or to other therapeutic options (approved or investigational) with documented evidence of clinical activity.

E3. For patients under chemotherapy /Immunotherapy/ biological- or targeted- or any other type of therapy + ICI before inclusion: Persistence of CTCAE ≥ Grade 2 toxicity due to prior combined agent (except alopecia (any grades), blood tests values according to inclusion criteria).

E4. Patient with any history of CTCAE Grade 4 irAEs under anti-PD-1/PD-L1 treatment or any history of CTCAE Grade 3 requiring steroid treatment (>10 mg/day prednisone or equivalent dose) for >12 weeks or CTCAE Grade 2 pneumonitis regardless of steroid treatment.

E5. History of severe (≥ Grade 3) allergic anaphylactic reactions to one of the components of NP137, standard ICI, premedication and/or any of their excipients.

E6. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.

E7. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years.

Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.

E8. Prior therapy or needs to be treated with a forbidden concomitant/concurrent therapies/procedures including:

* Any investigational agent or have used an investigational device. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 2 weeks or 5* ½ whichever is shorter after the last dose of the previous investigational agent.
* Radiotherapy within 4 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.Palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease and on non-target lesion is allowed.
* Major surgery within 4 weeks of start of study treatment. Participants must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment, C1D1.
* Anti-cancer treatment other than those specified in the protocol i.e. standard anti-PD1/PDL1
* Live or live-attenuated vaccine within 30 days prior to the first dose of study treatments. Note: killed are allowed.
* Immunosuppressive medication within 2 weeks with the exceptions of intranasal, topical and inhaled corticosteroids or systemic corticosteroids at doses which are not to exceed 10 mg/day of prednisone, or equivalent doses of another corticosteroid.

E9. Have a history of autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.

History of autoimmune disease which include but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis with the following exceptions:

* patients with a history of autoimmune-related hypothyroidism who are on stable thyroid replacement hormone therapy,
* patients with controlled Type 1 diabetes mellitus,
* patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are eligible provided that they meet the following conditions:

  * Rash must cover less than 10% of body surface area (BSA).
  * Disease is well controlled at baseline and only requiring low potency topical steroids.
  * No acute exacerbations of underlying condition within the previous 12 months requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoid, biologic agents, oral calcineurin inhibitors, high potency or oral steroids.

E10. Patients with HIV, active B or C hepatitis infection. Notes: Active hepatitis B i.e. chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening before C1D1. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. HBV DNA test must be performed in these patients prior to C1D1. Patients with a positive HBcAb test must have a negative HBV DNA test at screening. Active hepatitis C i.e. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA at screening.

E11. Patients with active tuberculosis. E12. Prior allogeneic bone marrow transplantation or solid organ transplant for another malignancy in the past.

E13. History of idiopathic pulmonary fibrosis, non-infectious pneumonitis/ interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease, drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan.

E14. Have an active infection requiring systemic therapy. E15. Pregnant or breastfeeding women. A WOCBP who has a positive urine pregnancy test (e.g. within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

E16. Patients placed under a legal protection regimen: Judicial Safeguards, curatorship or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-11-24 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR-12W) | 12 weeks
  Cohort 1 (SD): rate of patients with CR or PR according to RECIST V1.1 after the first 12 weeks of the NP137 as add on therapy.
Progression Free Rate at 12 weeks (PFR-12W) | 12 weeks
  Cohort 2 & 3 (primary and secondary refractory refractory): defined as the proportion of patients without documented disease progression according to RECIST V1.1 or documented clinical disease progression after the first 12 weeks of the NP137 as add on therapy.

SECONDARY OUTCOMES:
Objective Response Rate (ORR-12W) | 12 weeks
  Cohort 2 & 3: defined as the rate of patients with CR or PR according to RECIST V1.1 after the first 12 weeks of the NP137 as add on therapy
Time to objective response (ToR) | Every 12 weeks, up to 52 weeks
  All cohorts: defined as the time from C1D1 to the first documented and confirmed objective response as per RECIST V1.1
Duration of Response (DoR) | Every 12 weeks, up to 52 weeks
  All cohorts: defined as the time interval from the date of first occurrence of a documented objective response (CR or PR, whichever status is recorded first) until the first date that disease progression or death is documented, whichever occurs first. DOR will be assessed in patients who had an objective response. Patients who have not progressed and who have not died at the time of analysis will be censored at the time of last tumor assessment. If no tumor assessments were performed after the date of the first occurrence of a documented CR or PR, DOR will be censored at the date of the first occurrence of a documented CR or PR plus 1 day. DoR will be analysed using central read tumor assessments
Safety profile | from the date of first intake of study drug until 90 days after study drug discontinuation or at time of initiation of a new anti-cancer treatment
  any AEs graded using Common Terminology Criteria for Adverse Events (CTCAE) V5.0.

OTHER OUTCOMES:
Epithelial-mesenchymal transition (EMT) score evolution under treatment | before first adminitration of NP137, then after 6 weeks of treatment and in case of relapse
  Measurement of the EMT score under treatment on pre and on- treatment tumor biopsies
Modulation of the tumoral microenvironment | before first adminitration of NP137, then after 6 weeks of treatment and in case of relapse
  Evolution of tumor immune cells by multi-IF under treatment on pre and on-treatment tumor biopsies
Netrin-1 and UNC5B expression | before first adminitration of NP137, then, after 6 weeks of treatment and in case of relapse
  Netrin-1 and UNC5B expression by IHC on pre and on-treatment tumor biopsies and correlation between the variation of the Netrin-1/ UNC5B expression and the clinical response.
Gene expression and gene signature (RNAseq) | before first adminitration of NP137, then, after 6 weeks of treatment and in case of relapse
  Gene expression and gene signature (RNAseq) on pre and on-treatment tumor biopsies

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut de Cancérologie Strasbourg Europe (ICANS), Strasbourg
  - Institut Claudius Regaud (IUCT Oncopole), Toulouse